CLINICAL TRIAL: NCT02762630
Title: Use of a Novel Weight Bearing Cone Beam Computed Tomography (CBCT) Scanner for Imaging of the Patellofemoral Joint
Acronym: NPF
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, John Marzo, Associate Professor of Clinical Orthopedics, State University of New York at Buffalo
Other Study IDs: STUDY00000568
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Patellofemoral Joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Carestream Health Inc. weight bearing cone beam CT scanner

SUMMARY:
Healthy volunteers will have a weight bearing cone beam CT scan of their knee to assess normal alignment of the knee joint

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Be 16 or more years of age
* Subject is able to be positioned properly in the investigational device and be still during the exam to reduce the potential of motion during the images

Exclusion Criteria:

* Have a history of patella instability
* Have had any type of previous knee surgery
* Have had a significant fracture of the patellofemoral joint
* Have a knee ligament injury
* Are pregnant at the time of screening or become pregnant during the study
* Have a history of high radiation exposure (i.e., undergone radiation therapy)
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Tibial tubercle-trochlear groove (TT-TG) offset distance (mm) | 1 day